CLINICAL TRIAL: NCT07225296
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending Dose, Multiple Ascending Dose, and Food-effect Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GNS-3545 in Healthy Adult Subjects
Brief Title: A Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GNS-3545 in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genosco Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GNS-3545-P101
Record Dates: First submitted 2025-10-28; First posted 2025-11-06 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Intervention Model Description: This is a first-in-human, single ascending dose (SAD, Part 1) and multiple ascending dose (MAD, Part 2) study of orally administered GNS-3545 in healthy adults. Each cohort will include 8 participants (6 active, 2 placebo).
  In Part 1, a single oral dose will be administered under fasting conditions. In Part 2, once-daily dosing will be administered for 14 consecutive days under fasting conditions. Sequential cohorts will receive increasing doses, with dose escalation decisions based on safety and tolerability reviews by the Safety Review Committee (SRC). Six (6) cohorts (S1 to S6) are planned for evaluation in Part 1 (SAD), and Three (3) cohorts (M1 to M3) are planned for evaluation in Part 2 (MAD).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Parts 1 (SAD) and 2 (MAD) of the study will be conducted in a double-blind manner, in which both participants and investigators will be blinded to treatment assignment (active or placebo). Each cohort will include eight subjects randomized in a 3:1 ratio (six active and two placebo).
  The randomization code will be generated by a designated individual under the supervision of a statistician. All site and sponsor personnel involved in the study, except for the pharmacist (or designee) preparing study medication, will remain blinded.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GNS-3545 (Experimental): Part 1 (SAD): Six participants will be randomized to receive a single dose of GNS-3545 at the assigned dose level, while two participants will receive matching placebo.
  Part 2 (MAD): Six participants will be randomized to receive multiple doses of GNS-3545 at the assigned dose level once daily for 14 consecutive days, while two participants will receive matching placebo.
  Interventions: Drug: GNS-3545
- GNS-3545 Placebo (Placebo Comparator): Part 1 (SAD): Six participants will be randomized to receive a single dose of GNS-3545 at the assigned dose level, while two participants will receive matching placebo.
  Part 2 (MAD): Six participants will be randomized to receive multiple doses of GNS-3545 at the assigned dose level once daily for 14 consecutive days, while two participants will receive matching placebo.
  Interventions: Drug: GNS-3545 Placebo

INTERVENTIONS:
Drug: GNS-3545 — GNS-3545 will be administered as oral tablets at assigned dose levels to six of the eight participants within each cohort in Part 1 (SAD) and Part 2 (MAD).
  In Part 1, participants will receive a single dose on one occasion (Day 1). In Part 2, participants will receive daily dosing for 14 consecutive days.
  Arms: GNS-3545
Drug: GNS-3545 Placebo — The placebo will be administered as oral tablets identical in appearance to the GNS-3545 tablets to two of the eight participants within each cohort in Part 1 (SAD) and Part 2 (MAD).
  In Part 1, participants will receive a single placebo dose on one occasion (Day 1).
  In Part 2, participants will receive once-daily placebo doses for 14 consecutive days.
  Arms: GNS-3545 Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled Phase 1 study of SAD (Part 1) and MAD (Part 2) of orally administered GNS-3545 in healthy adult subjects. The food effect will be assessed in one cohort in Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female (of non-childbearing potential only), 18-55 years of age
* Male subjects must follow protocol specified contraception guidance
* Continuous non-smoker who has not used nicotine-containing products for at least 3 months prior to the first dosing
* BMI ≥ 18.0 and ≤ 32.0 kg/m2 at the screening visit and body weight of ≥ 50 kg
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, or vital signs, as deemed by the PI or designee
* No ECG findings of clinical significance as judged by the PI or qualified designee
* Understands the study procedures in the ICF and be willing and able to comply with the protocol

Exclusion Criteria:

* Is mentally or legally incapacitated or has significant emotional problems
* History or presence of clinically significant medical or psychiatric conditions
* History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study
* Surgical procedure or Administration of a live vaccination within 30 days prior to the first dose of the study drug
* History or presence of alcohol or drug abuse within the past 2 years prior to the first dosing
* History or presence of hepatic impairment
* History or presence of significant cardiovascular conditions or risk factors
* Subjects with a higher risk of adverse events in the setting of blood pressure decreases
* History or presence of hypersensitivity to compounds related to the study drug excipients
* Allergy to non-latex band aids, adhesive dressing, or medical tape
* Female subjects of childbearing potential or Female subject with a positive pregnancy test or who is lactating
* Positive urine drug or serum alcohol results
* Positive results at the screening visit for HIV, HBsAg, or HCV, or a clinically significant history of infection within 3 months prior to screening
* Inability or unwillingness to avoid use of medications, supplements, or substances that may affect CYP enzymes, drug transporters, blood pressure, or QT/QTc interval within the specified washout periods prior to dosing
* Has been on a diet incompatible with the on-study diet, or unable to swallow multiple tablets by mouth
* Has donated or lost more than 500 mL of blood within 56 days prior to the first dosing, or Plasma donation within 7 days prior to the first dosing
* Subjects with dietary restrictions that would prevent subjects from consuming a high-fat/high-calorie meal
* Participation in another clinical study within 30 days or 5 half-lives of the product prior to the first dosing
* Any reason determined by the PI or designee, in their opinion, that would prevent the subject's participation in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2026-06-12 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events (TEAEs) | Collection of TEAEs occurs from the point of first dose administration (Day 1 in each part) through to study completion (up to 8 days from the first dosing for Part 1 & up to 8 days from the last dosing for Part 2).
  Number and severity of treatment-emergent adverse events (TEAEs) following single and multiple doses of GNS-3545 and placebo

SECONDARY OUTCOMES:
Area under the time-concentration curve (AUC) from zero (pre-dose) to 24 hours (h) post-dose sample [0-24 h]) | Up to 4 days from the last dosing for Part 1 (SAD), Up to 4 days from the last dosing for Food Effect Cohort (Part 1), Up to 17 days from the last dosing for Part 2 (MAD)
  Pharmacokinetic profile of GNS-3545 and its active metabolite in plasma
Area under the time-concentration curve (AUC) from zero (pre-dose) to the time of the last measurable concentration (t) [0-t]) | Up to 4 days from the last dosing for Part 1 (SAD), Up to 4 days from the last dosing for Food Effect Cohort (Part 1), Up to 17 days from the last dosing for Part 2 (MAD)
  Pharmacokinetic profile of GNS-3545 and its active metabolite in plasma
Maximum observed concentration (Cmax) after a single dose and at steady state (Cmax,ss) | Cmax for up to 4 days from the last dosing for Part 1 (SAD), Cmax for up to 4 days from the last dosing for Food Effect Cohort (Part 1), Cmax & Cmax,ss up to 17 days from the last dosing for Part 2 (MAD)
  Pharmacokinetic profile of GNS-3545 and its active metabolite in plasma
Time to reach maximum observed concentration (Tmax) after a single dose and at steady state (Tmax,ss) | Tmax up to 4 days from the last dosing for Part 1 (SAD), Tmax for up to 4 days from the last dosing for Food Effect Cohort (Part 1), Tmax & Tmax,ss up to 17 days from the last dosing for Part 2 (MAD)
  Pharmacokinetic profile of GNS-3545 and its active metabolite in plasma
Cumulative amount excreted in urine over the collection interval (CumAe) after a single dose and at steady state (CumAe,ss) | CumAe for up to 4 days from the last dosing for Part 1 (SAD), CumAe,ss up to 17 days from the last dosing for Part 2 (MAD)
  Pharmacokinetic profile of GNS-3545 and its active metabolite in urine
Lag time before the first measurable concentration (Tlag) | Up to 4 days from the last dosing for Food Effect Cohort Only (Part 1)
  Pharmacokinetic profile of GNS-3545 and its active metabolite in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaron CPC, Inc., Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
At this stage, it is not planned that any IPD information will be shared.